CLINICAL TRIAL: NCT00466869
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Examine the Effect of Betahistine on Plasma Lipids in Patients Treated With Simvastatin
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: OBEcure Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BET203
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2007-08

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Betahistine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Betahistine

SUMMARY:
This is a randomized, double-blind, placebo-controlled, two-to three center study. The study will consist of 2 treatment groups (Betahistine 48 mg/day or matching placebo). Approximately 30 subjects (15 per treatment group) will be randomized into this 6-week study.

A single blinded placebo treated period of up to 14 days will be used to determine subjects suitability for inclusion in the trial.

In order that a patient will be defined as valid for inclusion in the study, patients should be able to present consistent LDL-C values, taken prior to randomization (at screening visit 1 and screening visit 2), without deviation of more than 12% of each value from their mean.

Within one week from the second screening visit, subjects who meet all inclusion criteria and none of the exclusion criteria will be randomly assigned to 1 of the following treatment groups:

* Betahistine 24 mg BID (48 mg/day total), or
* Matching placebo BID.

Double-blind treatment will continue for 4 weeks. Study medication (betahistine and/or matching placebo) will be administered BID (before lunch and before dinner).

During the study, subjects will undergo dietary assessment.

The primary efficacy parameter is change in LDL-C from baseline (randomization) to Week 4 and the percentage of patients that reduce their LDL-C by 10% or more.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent;
* Male or female subjects 30 to 75 years of age;
* Treated with Simvastatin (Simovil,C500,Simvacor,Simvastatin-Teva,Simvaxon)in dose that does not exceed 40 mg/day.
* Has been on a stable (unchanged) dose of Simvastatin for at least 3 months prior to screening;
* If female, is nonlactating, has a negative urine pregnancy test result, and does not plan on becoming pregnant during the study, or not of childbearing potential (hysterectomy or tubal ligation at least 6 months prior to randomization or post-menopausal for 1 year); if of childbearing potential (including peri-menopausal women who have had a menstrual period within one year) must practice or be willing to continue to practice appropriate birth control (such as implants, injectables, oral contraceptives, some intrauterine contraceptive devices, sexual abstinence, tubal ligation, or a vasectomized partner) during the entire study duration
* Consistent LDL-cholesterol values, taken at Visit 1 and 2 (screening visit 1 and screening visit 2), without deviations of more than 12% of each value from their mean.
* Patients should keep a stable diet and constant exercise activities during the last 3 months, as per the patients statements.
* Patients are compliant (taking > 80%) with study medication during the screening period.

Exclusion Criteria:

* Has uncontrolled hyperlipidemia (triglycerides [TG] >=300mg/dL or low-density lipoprotein cholesterol [LDL-C] >160 mg/dL or < 100mg/dL
* Has recently started or plans on starting a smoking cessation program;
* Has a BMI of less than 18.5 kg/m2 or higher than 40 kg/m2
* Has had a major change in daily physical activity (e.g., initiation of an exercise program) or started a weight loss program within 90 days prior to screening;
* Is unwilling or unable to participate in a dietary assessment as part of the study;
* Has a clinically significant history or presence of any of the following conditions:

  * History of myocardial infarction, cerebrovascular accident, stroke, unstable angina , percutaneous transluminal coronary angioplasty (PTCA), coronary artery bypass graft (CABG), cardiac valve abnormalities that requires the use of anticoagulants or SBE prophylaxis, within the six months prior to the screening visit 1.
  * Congestive heart failure (NYHA class 3 or 4).
  * Significant arrhythmia or conduction disturbances (e.g.: second or third degree AV block without a cardiac pacemaker, multiple multifocal ventricular ectopic beats).
  * History of pancreatitis and/or serum amylase >2xULN) in addition to clinical signs of pancreatitis.
  * History of gastro-intestinal disease (e.g. Crohn's disease) which could result in impaired absorption of the study drug.
  * Type 1 diabetes mellitus;
  * Treated Type 2 diabetes mellitus ( metformin monotherapy and/or diet are allowed ) with HbA1c >8%;
  * Severe type 2 diabetes with history of ketoacidosis or diabetic ulcers, or presence of retinopathy, neuropathy, or nephropathy;
  * Renal insufficiency defined as a serum creatinine>=1.5 mg/dL (133 µmol/L) at screening;
  * Previous malignant disease within 5 years of screening: (except cervical carcinoma in situ, adequately treated basal cell carcinoma, or superficial bladder tumors [Ta, Tis & T1]
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2 x ULN;
  * CPK (creatine phosphokinase) >3 x ULN
  * Hypothyroid patient defined as: TSH > 7.5 mU/l or 5<TSH <7.5 mU/l and total T4< 4.00 mcg/dl (51.5 nmol/l) (regardless if the patient is on replacement therapy or not).
  * Plans on having any surgery (elective or otherwise) during the course of the study;
  * Has uncontrolled hypertension (sitting blood pressure > 160/100 mmHg at screening or randomization).
  * History of asthma;
  * History of peptic ulcers;
  * History of HIV
  * Any other disease or condition which might preclude the patient's regular participation to the study (e.g. other endocrine diseases, acute or chronic infections, known or suspected drug or alcohol abuse or has psychiatric or neurological disorders requiring chronic medications (e.g., antidepressants);
  * Chronic or as needed use of antihistamines;
* Has not been on a stable treatment regimen with any of the following medications for a minimum of 90 days prior to screening:
* Hormone replacement therapy;
* Oral contraceptives;
* Antihypertensive agents;
* Metformin;
* hyroid replacement therapy;
* Has been treated over the past 60 days, is currently treated, or is expected to require or undergo treatment with any of the following excluded medications:
* All prescription or over-the-counter agents taken for the purpose of treating dyslipidemia, including (but not limited to) the following agents:

  * Statins such as Rosuvastatin (Crestor), Fluvastatin (Lescol), Atorvastatin (Lipitor ,Torid), Pravastatin (Pravalip, Pravastatin).
  * Fibrates such as Bezafibrate (Bezafibrate 400 Sr,Norlip) Ciprofibrate Lipanor)
  * Bile acid sequestrant such as Colestipol (Colestid)
  * Cholesterol absorption inhibitor such as Ezetimibe (Ezetrol)
  * Nicotinic acid derivative such as Acipimox (Olbetam)
  * Omega-3-acid such as Triomar, Omacor
  * Over-the-counter hypolipidemic agents (e.g., vitamins, herbal supplements or other alternative remedies);
* All prescription or over-the-counter agents taken for the purpose of weight reduction, including (but not limited to) the following anti obesity agents:
* Prescription drugs such as orlistat (Xenical®), sibutramine (Reductil), and phentermine (Razin).
* Psychotropic/neurological agents including the following:
* Antipsychotic agents (e.g., Olanzapine, Clozapine, Risperidol, Lithium, etc.).
* Antiepileptic agents (e.g., Topamax®, Zonegran®, valproate, carbamazepine).
* Antidepressant agents including the following: monoamine oxidase inhibitors, bupropion (Zyban®), tricyclic antidepressants, and tetracyclic antidepressants; and selective serotonin reuptake inhibitors (e.g., Prozac®, Paxil®, Zoloft®, etc.);
* Systemic steroids administered by oral, intravenous, or intramuscular route;
* Drugs that directly affect gastrointestinal motility (e.g., Reglan® and Propulsid®, and chronic [taken for more than 10 days within a 6-month period prior to screening visit 1] macrolide antibiotics such as erythromycin and newer derivatives):
* Calcitonin (e.g., Miacalcin®);
* Insulin;
* α-glucosidase inhibitor (Prandase®);
* Sulfonylureas (e.g., Amaryl®, Diabitex®, Glibetic®, Gluben®, Gluco- Rite® Novonorm® Orsinon®); Or
* Meglitinide (e.g. NovoNorm)
* Rosilitazone (e.g. Avandamet ® Avandia® Rossini®)
* Receipt of any investigational treatment (drug or device) within 30 days prior to screening;
* Is an immediate family member of personnel directly affiliated with the study at the investigative site, or is personally directly affiliated with the study at the investigative site; or
* Is employed by OBEcure Ltd.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-05; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary efficacy parameter is change in LDL-C from baseline (randomization) to Week 4 and the percentage of patients that reduce their LDL-C by 10% or more.

SECONDARY OUTCOMES:
Change in Total Cholesterol from baseline (randomization) to Week 4.
Change in Triglycerides l from baseline (randomization) to Week 4.
Change in High density lipoprotein (HDL-C) from baseline (randomization) to Week 4.
Change in Total cholesterol to HDL-C ratio from baseline (randomization) to Week 4.
Change in ApoB from baseline (randomization) to Week 4.
Change in hemoglobin A1c [HbA1c], and fasting plasma glucose [FPG] from baseline (randomization) to Week 4.
Change in Caloric intake and macronutrients intake from baseline (randomization) to Week 4.
Change in body weight from baseline (randomization) to Week 4.
Change in waist circumference from baseline (randomization) to Week 4.

CONTACTS AND LOCATIONS:
Overall Officials: Yaffa Beck, Dr., Study Chair
Locations (2):
- Israel (2):
  - Internal Medicine Department A-Wolfson Medical Center, Holon
  - Internal Medicine Department A-Meir Medical Center, Kfar Saba